CLINICAL TRIAL: NCT03649750
Title: A Phase I, Open-label, Single-dose, Randomized, 2-way Cross-over Study Designed to Examine the Relative Bioavailability of Guaifenesin When a Mucinex Extended Release 600 mg Bi-layer Tablet is Taken Under Fasted Compared to Fed Conditions in Normal Healthy Volunteers
Brief Title: Mucinex® ER 600 mg Bi-Layer Tablet Fed and Fasted
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-MUC-01
Record Dates: First submitted 2018-08-20; First posted 2018-08-28 (Actual); Results first posted 2019-02-22 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Acetylcysteine; Guaifenesin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: Mucinex® 600 mg (fast) (Experimental): Mucinex® 600 mg ER bi-layer tablet by mouth after 10 hours fasting and subject will fast at least 4 hours post-dose
  Interventions: Drug: Mucinex®
- Treatment B: Mucinex® 600 mg (fed) (Experimental): Mucinex® 600 mg ER bi-layer tablet by mouth in fed condition. After an overnight fast of at least 10 hours, subjects will consume a high fat, high calorie breakfast starting 30 minutes prior to drug administration
  Interventions: Drug: Mucinex®

INTERVENTIONS:
Drug: Mucinex® — Mucinex® 600 mg ER bi-layer tablets
  Other Names: guaifenesin

SUMMARY:
Determine and compare the plasma concentrations of Mucinex® Extended Release (ER) 600 mg bi-layer tablet in normal healthy volunteers in fed and fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent was obtained (i.e. be informed of the nature of the study and given written consent prior to any study procedure). Able to read, understand, and sign the informed consent, after the nature of the study had been explained.
2. Age: 18 to 55 years of age, inclusive.
3. Sex: male or female.
4. Status: Healthy subjects.
5. BMI: ≥18.0 and ≤28.0 kg/m2.
6. No clinically significant findings in vital signs measurements at screening.
7. No clinically significant abnormal laboratory values at screening.
8. No clinically significant findings from a 12-lead electrocardiogram (ECG) at screening.
9. Had no significant diseases or clinically relevant medical condition in the opinion of the Investigator
10. Males who participated in this study were willing to:

    * remain abstinent [not engage in sexual intercourse] from the start of drug administration until 90 days after the end of the study or
    * used (or their partner used, as applicable) two effective methods of birth control [condom, diaphragm, cervical cap, vaginal sponge, spermicide, IUD, tubal ligation, vasectomy, or hormonal contraceptives] from the start of drug administration until 90 days after the end of the study.

    Females who participated in this study were:
    * unable to have children (e.g., post-menopausal, hysterectomy);
    * willing to remain abstinent [not engage in sexual intercourse] from 21 days prior to drug administration until 30 days after the end of the study; or
    * willing to use two effective methods of birth control [condom, diaphragm, cervical cap, vaginal sponge, spermicide, non-hormonal Intrauterine Device (IUD) (in place for 3 months), tubal ligation, partner has vasectomy, hormonal contraceptives for 3 months prior to drug administration] from 30 days prior to drug administration until 30 days after the end of the study.
11. Had no clinically significant findings from a physical examination.

Exclusion Criteria:

1. Employee of Pharma Medica Research Inc. (PMRI) or Reckitt Benckiser.
2. Partner or first-degree relative of any Investigator at PMRI.
3. Known history or presence of any clinically significant medical condition.
4. Known or suspected carcinoma.
5. Presence of hepatic or renal dysfunction.
6. Presence of clinically significant gastrointestinal disease or history of malabsorption within the year preceding the study.
7. Known history or presence of galactose or fructose intolerance, sucrase-isomaltase insufficiency, Lapp lactase insufficiency, galactosemia, or glucose-galactose malabsorption syndrome.
8. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
9. History of drug or alcohol or medicinal product addiction requiring treatment within the two years preceding the study or excessive alcohol consumption (more than 10 units per week)

   Note: one unit is defined as 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of spirits.
10. Positive test result for serum Human Chorionic Gonadotropin (hCG) consistent with pregnancy (females only), HIV, Hepatitis B surface antigen or Hepatitis C antibody.
11. Positive test result for urine drugs of abuse (cannabinoids, opiates, amphetamines, cocaine, phencyclidine, tricyclic antidepressants, barbiturates, methadone and benzodiazepines) or urine cotinine.
12. Difficulty fasting or consuming standard meals.
13. Females who were lactating.
14. Did not tolerate venipuncture.
15. Use of tobacco or nicotine-containing products within 12 months prior to drug administration.
16. On a special diet within 30 days prior to drug administration (e.g., liquid, protein, raw food diet).
17. Donation or loss of whole blood (including clinical trials):

    * ≥50 ml and ≤499 ml within 30 days prior to drug administration
    * ≥500 ml within 56 days prior to drug administration
18. Females who had started taking hormonal contraceptives or had changed their method or brand of hormonal birth control within 3 months prior to drug administration.
19. Had a tattoo or body piercing within 30 days prior to drug administration.
20. Use of drugs of the monoamine oxidase inhibitor (MAOI) class within 30 days prior to drug administration.
21. Known history or presence of hypersensitivity, intolerance or idiosyncratic reaction to guaifenesin or any other drug substances with similar activity.
22. Previously enrolled in this study.
23. Participated in another clinical trial or received an investigational product within 30 days prior to drug administration.
24. Unable in the opinion of the Investigator to comply fully with the study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-05-29 (Actual); Primary Completion 2013-08-07 (Actual); Study Completion 2013-08-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-centre study.
Pre-assignment Details: Total Thirty-six (36) subjects were enrolled in the study among them 36 subjects completed the study.
Groups:
- Cohort 1(Mucinex Fed or Mucinex Fast in Period 1 and Period 2): Treatment A (Test): Single dose Mucinex® 600 mg Extended Release bi-layer tablet by mouth under overnight fasting.
  Treatment B (Test): Single dose Mucinex® 600 mg Extended Release bi-layer tablet by mouth under high calorie breakfast fed.
  Cohort 1
  Period 1 - Treatment A or Treatment B at Sequence AB.
  Period 2 - Treatment B or Treatment A at Sequence BA.
  Scheduled Washout of 7 days between drug doses.
- Cohort 2(Mucinex Fast or Mucinex Fed in Period 1 and Period 2): Treatment A (Test): Single dose Mucinex® 600 mg Extended Release bi-layer tablet by mouth under overnight fasting.
  Treatment B (Test): Single dose Mucinex® 600 mg Extended Release bi-layer tablet by mouth under high calorie breakfast fed.
  Cohort 2
  Period 1 - Treatment A or Treatment B at Sequence AB.
  Period 2 - Treatment B or Treatment A at Sequence BA.
  Scheduled Washout of 7 days between drug doses.
Period: Period 1
Arm/Group | Cohort 1(Mucinex Fed or Mucinex Fast in Period 1 and Period 2) | Cohort 2(Mucinex Fast or Mucinex Fed in Period 1 and Period 2)
Started | 12 | 24
Completed | 12 | 24
Not Completed | 0 | 0
Period: Washout: 7 Days
Arm/Group | Cohort 1(Mucinex Fed or Mucinex Fast in Period 1 and Period 2) | Cohort 2(Mucinex Fast or Mucinex Fed in Period 1 and Period 2)
Started | 12 | 24
Completed | 12 | 24
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Cohort 1(Mucinex Fed or Mucinex Fast in Period 1 and Period 2) | Cohort 2(Mucinex Fast or Mucinex Fed in Period 1 and Period 2)
Started | 12 | 24
Completed | 12 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pharmacokinetic (PK) Dataset Subjects from whom the observation/estimation of Cmax and AUC measures/parameters were possible for two periods were included in the PK dataset.
Groups:
- Pharmacokinetic (PK) Dataset: Treatment A (Test): Single dose Mucinex® 600 mg Extended Release bi-layer tablet by mouth under overnight fasting.
  Treatment B (Test): Single dose Mucinex® 600 mg Extended Release bi-layer tablet by mouth under high calorie breakfast fed.
  Cohort 1
  Period 1 - Treatment A or Treatment B at Sequence AB.
  Period 2 - Treatment B or Treatment A at Sequence BA.
  Scheduled Washout of 7 days between drug doses.
  Cohort 2
  Period 1 - Treatment A or Treatment B at Sequence AB.
  Period 2 - Treatment B or Treatment A at Sequence BA.
  Scheduled Washout of 7 days between drug doses.
Arm/Group | Pharmacokinetic (PK) Dataset
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19
Height [Mean (Standard Deviation); unit: cm] | 170.8 (10.1)
Weight [Mean (Standard Deviation); unit: kg] | 72.3 (10.4)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 24.7 (2.1)
Age [Number; unit: participants]
  18 - 40 years | 21
  41 - 64 years | 15
Race [Number; unit: participants]
  Asian | 6
  Black or African American | 8
  White | 22

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Guaifenesin
Description: Maximum measured analyte concentration over the sampling period.
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 9, 10, 11, 12, 14, 16, 20, and 24 hours (Period 1 and 2)
Population: Pharmacokinetic (PK) Dataset are the Subjects from whom the observation/estimation of Cmax and AUC measures/parameters will be possible for two periods will be included in the PK dataset.
  The PK dataset will be defined prior to the assay of samples.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Treatment A: Mucinex® 600 mg (Fast): Single dose Mucinex® 600 mg Extended Release bi-layer tablet by mouth under overnight fasting.
- Treatment B: Mucinex® 600 mg (Fed): Single dose Mucinex® 600 mg Extended Release bi-layer tablet by mouth under high calorie breakfast fed.
Arm/Group | Treatment A: Mucinex® 600 mg (Fast) | Treatment B: Mucinex® 600 mg (Fed)
Number analyzed (Participants) | 36 | 36
ng/ml | 1066.11 (429.91) | 1117.31 (424.82)

2. Primary Outcome: Area Under Plasma Concentration-time Curve From Time 0 to the Last Measurable Plasma Concentration (AUCt) of Guaifenesin
Description: The area under the analyte concentration versus time curve, from time zero (0) to the time of the last measurable analyte concentration (t), as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Population: Pharmacokinetic Dataset
Measure: Mean (Standard Deviation); unit: ng·h/ml
Arm/Group | Treatment A: Mucinex® 600 mg (Fast) | Treatment B: Mucinex® 600 mg (Fed)
Number analyzed (Participants) | 36 | 36
ng·h/ml | 4052.10 (1495.48) | 4084.90 (1380.20)

3. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Guaifenesin
Description: Time of the maximum measured analyte concentration over the sampling period.
Time Frame: as for outcome 1
Population: Pharmacokinetic Dataset
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment A: Mucinex® 600 mg (Fast) | Treatment B: Mucinex® 600 mg (Fed)
Number analyzed (Participants) | 36 | 36
h | 0.68 (0.32) | 3.33 (1.36)

4. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time 0 to Infinity (AUCinf) of Guaifenesin
Description: The area under the analyte concentration versus time curve from time zero to infinity.
  AUCinf = AUCt + Cp/Kel,
  where Cp is the predicted analyte concentration at the time of the last measurable analyte concentration.
Time Frame: as for outcome 1
Population: Pharmacokinetic Dataset
Measure: Mean (Standard Deviation); unit: ng·h/ml
Arm/Group | Treatment A: Mucinex® 600 mg (Fast) | Treatment B: Mucinex® 600 mg (Fed)
Number analyzed (Participants) | 36 | 36
ng·h/ml | 4104.47 (1555.87) | 4092.53 (1382.77)

5. Secondary Outcome: Terminal Elimination Rate Constant (Kel) of Guaifenesin
Description: Elimination rate constant calculated from the slope of the terminal portion of the plasma profile calculated by least-squares regression of log (concentration) versus time.
Time Frame: as for outcome 1
Population: Pharmacokinetic Dataset
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Treatment A: Mucinex® 600 mg (Fast) | Treatment B: Mucinex® 600 mg (Fed)
Number analyzed (Participants) | 36 | 36
1/h | 0.3862 (0.1717) | 0.6788 (0.1343)

6. Secondary Outcome: Terminal Elimination Half-life (T½) of Guaifenesin
Description: Terminal elimination half-life, calculated from the equation: thalf = In(2)/Kel.
Time Frame: as for outcome 1
Population: Pharmacokinetic Dataset
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Treatment A: Mucinex® 600 mg (Fast) | Treatment B: Mucinex® 600 mg (Fed)
Number analyzed (Participants) | 36 | 36
h | 2.46 (2.62) | 1.07 (0.29)

7. Secondary Outcome: Relative Bioavailability (RF) of Guaifenesin
Description: Relative bioavailability for each formulation will be defined as:
  (AUC0-inf Fasting ÷ AUC0-inf Fed) x (Fed dose ÷ Fasting dose)
Time Frame: as for outcome 1
Population: Outcome involved analyzing data from both intervention groups (Fed and Fasting) in combination as per the provided formula, therefore, separate analysis for each intervention cannot be reported
Measure: Mean (Standard Deviation); unit: Percent bioavailability
Groups:
- All Study Participants: Single dose Mucinex® 600 mg Extended Release bi-layer tablet by mouth under overnight fasting and fed.
Arm/Group | All Study Participants
Number analyzed (Participants) | 36
Percent bioavailability | 1.0081 (0.1655)

8. Secondary Outcome: Number of Adverse Events(AEs) Experienced by Participants
Description: Intensity determination Mild=AE does not limit usual activities;subject may experience slight discomfort Moderate=AE results in some limitation of usual activities;subject may experience significant discomfort Severe=AE results in an inability to carry out usual activities;subject may experience intolerable discomfort or pain Unassessable/Unclassifiable=Insufficient information to be able to make an assessment Conditional/Unclassified=Insufficient information to make an assessment at present(causality is conditional on additional information) Unrelated=No possibility that the AE was caused by study drug Unlikely=Slight but remote chance that the AE was caused by study drug but the balance of judgment is that it was most likely not due to the study drug Possible=Reasonable suspicion that the AE was caused by the study drug Probable=Most likely that the AE was caused by study drug Certain=The AE was definitely caused by study drug
Time Frame: Up to period 2 (8.3 days/200 hours)
Population: Pharmacokinetic Dataset
  Investigational Medicinal Product(IMP)
Measure: Number; unit: Events
Arm/Group | Treatment A: Mucinex® 600 mg (Fast) | Treatment B: Mucinex® 600 mg (Fed)
Number analyzed (Participants) | 36 | 36
Events
  TEAE by severity: Mild | 11 | 14
  TEAE by severity: Moderate | 0 | 0
  TEAE by severity: Severe | 0 | 0
  Relationship to IMP: Unassessable/Unclassifiable | 3 | 5
  Relationship to IMP: Conditional /Unclassified | 0 | 0
  Relationship to IMP: Unrelated | 2 | 0
  Relationship to IMP: Unlikely | 0 | 0
  Relationship to IMP: Possible | 6 | 9
  Relationship to IMP: Probable | 0 | 0
  Relationship to IMP: Certain | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 8.3 days/ (200 hours)
Arm/Group | Treatment A: Mucinex® 600 mg (Fast) | Treatment B: Mucinex® 600 mg (Fed)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 8/36 | 10/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Mucinex® 600 mg (Fast) (N=36) | Treatment B: Mucinex® 600 mg (Fed) (N=36)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1)
Vessel puncture site swelling (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 5 (5) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No